CLINICAL TRIAL: NCT00297349
Title: An Open-label Observation Study of Topiramate Administration as Adjuvant Therapy for Focal Epilepsy, Lennox-Gastaut Syndrome Epileptic Seizures and Generalized Tonoclonic Seizures in Adults and Children Aged 2 Years and Older
Brief Title: A Study of the Safety of Topiramate Given in Combination With Other Medications in Adults and Children With Seizures
Status: Completed | Type: Observational
Sponsor: Janssen Cilag Pharmaceutica S.A.C.I., Greece (Industry)
Responsible Party: Medical Affairs Director, Janssen Cilag Pharmaceutica S.A.C.I., Greece
Other Study IDs: CR003472
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Seizures; Epilepsy
Keywords: Seizures; Epilepsy; Tonic-clonic; Lennox-Gastaut Syndrome; Focal Epilepsy; Topiramate; Epilepsy in Children
MeSH Terms: conditions — Seizures; Epilepsy; Lennox Gastaut Syndrome; Epilepsies, Partial | interventions — Topiramate

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — Individualization of the treatment should begin from 25 mg for 1 week.

SUMMARY:
The purpose of this observational study is to evaluate the safety of topiramate when used in combination with other medications for seizures in adults and children.

DETAILED DESCRIPTION:
Topiramate is a medication that is approved for the treatment of seizures. In accordance with International guidelines, studies are conducted after a drug is marketed to continue to evaluate and expand the knowledge regarding its safety. This is an open-label, multi-center observational safety study to collect safety information for oral topiramate given in addition to other medications for 3 types of seizures in adults and in children aged 2 years and older.The 3 seizures types are focal epilepsy, LENNOX-GASTAUT syndrome epileptic seizures and generalized tonic-clonic seizures. Patients whose previous treatment for seizures (one or more antiepileptic drugs) has been judged by their physician to be non-satisfactory will receive 6 months of treatment with topiramate in addition to other antiepileptic medication as prescribed by their physician. Topiramate will be given at low doses initially and gradually increased as necessary to control seizure activity in accordance with Summary of Product Characteristics (SmPC). Patients will be asked to keep a diary of adverse events and seizure activity. Safety evaluations (incidence of adverse events, physical examinations, vital signs and laboratory tests) will be performed throughout the study per investigators usual standard of care. At the end of the study, the treating physician may continue treatment with topiramate and other medication as appropriate. The study hypothesis is that topiramate given in combination with other antiepileptic medications will be effective in achieving and maintaining control of seizure activity and is well-tolerated. 225 adult patients and children aged 2 years or older will be enrolled in the study. Study participants should demonstrate focal epilepsy or epileptic seizures of the LENNOX-GASTAUT syndrome or generalized tonoclonic seizures, who have undergone treatment with one or more antiepileptic drugs and whose treatment should be judged by the investigator as non-satisfactory. Observational study - No investigational drug administered.

ELIGIBILITY:
Inclusion Criteria:

* Non-premenopausal female patients using a medically acceptable contraceptive method as discussed with their doctor
* History of the type of seizure during the period prior to inclusion in the study and sufficient medical records to document this. Prior treatment until inclusion in the study with one or more antiepileptic drug treatment judged non-satisfactory by the investigator

Exclusion Criteria:

* Patients not suffering from epilepsy, whose seizures are due to other causes including disease, exposure to harmful substances, active infection or tumor
* Patients with a history of generalized status epilepticus (prolonged seizures) within the last three months
* Patients with progressive brain tumor or other progressive or degenerative disorders
* Patients with a history (within the previous six months) of mental or emotional disorders requiring shock treatment or major sedation, monoamine oxidase (MAO) inhibitors or medications which affect the central nervous system
* Patients with any medical or social condition that may affect their ability to take part in study or the safety of the study
* Patients who cannot take the drug or fill in the diary, either alone or with help. If help is needed, it should be permanently available throughout the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 225 adult patients and children aged 2 years or older will be enrolled in the study. Study participants should demonstrate focal epilepsy or epileptic seizures of the LENNOX-GASTAUT syndrome or generalized tonoclonic seizures, who should have undergone treatment with one or more antiepileptic drugs and whose treatment should be judged by the inverstigator as non-satisfactory.
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2003-11; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety of oral topiramate as adjuvant therapy for focal epilepsy, Lennox-Gastaut syndrome epileptic seizures and the generalized tonoclonic seizures in adults and children aged 2 years and older. | At visit 3-8

SECONDARY OUTCOMES:
Safety & tolerability evaluation will be performed by reporting AEs & Clinical labs. | Visits:3-8
Evaluation of efficacy will be performed with the aid of descriptive statistics. | Visits:3-8
Overall assessments of the improvement in the seriousness of seizures will be performed. | Visits:3-8

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pharmaceutica S.A.C.I. Clinical Trial, Study Director — Janssen-Cilag Pharmaceutica S.A.C.I.